CLINICAL TRIAL: NCT01020955
Title: Effects on Insulin Sensitivity and Body Composition of GH and IGF-I in Adult-GHD With Impaired Glucose Tolerance or Diabetes
Brief Title: Metabolic Effects of GH and IGF-I in Growth Hormone Deficient(GHD) and Diabetes and Impaired Glucose Tolerance(IGT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Hoeybye, MD, PhD, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: GH/IGF-I
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes
Keywords: GH and IGF-I; growth hormone deficiency and IGT or diabetes
MeSH Terms: conditions — Diabetes Mellitus; Dwarfism, Pituitary | interventions — mecasermin; Insulin-Like Growth Factor I

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NutropinAq and Increlex (Active Comparator): NutropinAq (0.15 mg/day for 1 month, 0.3 mg/day for 5 months) and Increlex (15 µg/kg/day for 1 month and 30 µg/kg/day for 5 months).
  Interventions: Drug: NutropinAq (GH) and Increlex (IGF-I)
- NutropinAq and placebo (Placebo Comparator): NutropinAq (0.15 mg/day for 1 month, 0.3 mg/day for 5 months) and placebo for 6 months.
  Interventions: Drug: NutropinAq and placebo

INTERVENTIONS:
Drug: NutropinAq (GH) and Increlex (IGF-I) — NutropinAq (GH)(0.15 mg/d for 1 month, 0.3 mg/d for 5 months) and Increlex (IGF-I) (15 µg/kg/d for 1 month, 30 µg/kg/d for 5 months)
  Other Names: NutropinAq (GH); Increlex (IGF-I)
  Arms: NutropinAq and Increlex
Drug: NutropinAq and placebo — NutropinAq (0.15 mg/d for 1 month, 0.3 mg/d for 5 months) and placebo for 6 months.
  Other Names: NutropinAq (GH); Placebo
  Arms: NutropinAq and placebo

SUMMARY:
The aim of this study is to measure effects of the combined treatment with GH and IGF-I on glucose sensitivity and body composition in patients with GHD and IGT or diabetes.

DETAILED DESCRIPTION:
The study was a 6 months randomised placebo controlled trial of adults with GHD and type 2 diabetes. All receive GH (0.15 mg/day for 1 month, 0.3 mg/day for 5 months) and are randomised to IGF-I or placebo (15 µg/kg/day for 1 month and 30 µg/kg/day for 5 months). Glucose metabolism is evaluated with euglycemic hyperinsulinemic clamp and body composition by computed tomography (CT) and bio impedance;.

ELIGIBILITY:
Inclusion Criteria:

1. Verified profound GH deficiency. If the patient is already on GH replacement therapy this must have been commenced at least 6 months prior to study entry.
2. Impaired glucose tolerance test or diabetes (stable on oral antidiabetic medication for at least 3 months)
3. HbA1C<7.5%
4. Age 18-70 years
5. Each patient must sign an informed consent document before inclusion in the study
6. Women of childbearing potential must provide a negative pregnancy test before study start, and they must agree to use an effective method of contraception such as double barrier contraception, an injectable or implanted hormonal contraceptive, combined oral contraceptive or an intra-uterine device (IUD). The patient must agree to continue to use the contraceptive for two weeks after the last injection of IMP. Women without childbearing potential are defined as being postmenopausal for at least 1 year, or permanently sterilised at least 3 months before study entry.

   -

Exclusion Criteria:

1. Known or suspected allergy to GH or IGF-I preparation
2. Insulin treatment
3. Proliferative retinopathy
4. Previous malignancy or other serious diseases (ex severe cardiovascular diseases, severe infections). Patients with a history of cancer can be included if they have been treated with curative therapy and have been disease free for more than 5 years. Patients with cardiac failure are not included.
5. Increased liver enzymes (ASAT or ALAT>2.5 normal range)
6. S-creatinine above 120 umol/L
7. Patients with active hyperthyroidism and untreated hypothyroidism
8. Pregnancy
9. Lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | start and 6 months

SECONDARY OUTCOMES:
body composition | start and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Hoeybye, MD, Principal Investigator — Karolinska UH
Locations (1):
- Department of Endocrinology, karolinska University hospital, Solna, Sweden, Sweden